CLINICAL TRIAL: NCT02123589
Title: The Psychological Effects of Different Sedation Protocol on Mechanically Ventilated Critically Ill adults-a Prospective, Randomized and Controlled Trial
Brief Title: The Psychological Effects of Different Sedation Protocol on Mechanically Ventilated Critically Ill Adults.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kangyan, Physician, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: West ChinaH Sedation
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Sedative Withdrawal Delirium
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deep sedation (Experimental): Injection of 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,then continuous intravenous infusion 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl to maintain sedation until attaining the target level of sedation,RASS score between -5 and -3
  Interventions: Drug: Deep sedation(midazolam and fentanyl )
- Deep and daily interruption of sedation (Experimental): Injection of 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,then continuous intravenous infusion 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl to maintain sedation until attaining the target level of sedation,RASS score between -5 and -3.and from the second day after subject was admitted in ICU, daily interruption of sedation will be taken .
  Interventions: Drug: Deep and daily interruption of sedation(midazolam and fentanyl )
- Light sedation (Experimental): Injection of 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,then continuous intravenous infusion 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl to maintain sedation until attaining the target level of sedation,RASS score between -2 and +1.
  Interventions: Drug: Light sedation(midazolam and fentanyl )

INTERVENTIONS:
Drug: Deep sedation(midazolam and fentanyl ) — 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,IV; 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl,continuous intravenous infusion ; the target level of sedation,RASS score between -5 and -3
  Arms: Deep sedation
Drug: Deep and daily interruption of sedation(midazolam and fentanyl ) — 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,IV; 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl continuous intravenous infusion ; The target level of sedation,RASS score between -5 and -3. Daily interruption of sedation will be taken from the second day after admitted in ICU
  Arms: Deep and daily interruption of sedation
Drug: Light sedation(midazolam and fentanyl ) — 0.05~0.1mg/kg midazolam and 1~2μg/kg fentanyl,IV; 0.05mg/kg.h midazolam and1~2μg/kg.h fentanyl,continuous intravenous infusion ; The target level of sedation,RASS score between -2 and +1;
  Arms: Light sedation

SUMMARY:
The study was designed to explore the effects of different sedation protocol on incidence rates of delirium and PTSD in severe patients with mechanically ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Critically ill adults whose expected time of mechanical ventilation is longer than 24 hours
* Aged between 18 years old to 85 years old.

Exclusion Criteria:

* Subjects with brain injury;
* History of cardiopulmonary resuscitation;
* Mental disability;
* Taken neuromuscular blocking drugs;
* Inability to exchange;
* Contraindicated to midazolam or morphine;
* Inconvenience to daily interruption

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The incident rate of delirium | From weaning to discharged from ICU,about 7 days.
The incident rates of PTSD | 30th day and 180th day after discharged from ICU
The duration of delirium | From weaning to discharged from ICU,about 7 days.

SECONDARY OUTCOMES:
Incidence rate of unexpected extubation | From intubation to weaning,about 7 days
Dosage of analgesics and sedatives | From intination of analgesics and sedatives to stopping drug appication,about 7 days
The duration of mechanical ventilation | From intubation to weaning,about 7days
Duration of ICU | From admitted to ICU to discharged from ICU,about 7 days
The whole hospitalization time | From admitted to hospital to discharged from hospital,about 7 days
Patients' death rates within ICU stay | From admitted to ICU to discharged from ICU,about 7 days
Patients' death rates within hospitalized stay | From admitted to hospital to discharged from hospital,about 7 days
The cost in ICU | From admitted to ICU to discharged from ICU,about 7 days
The total cost in hospital | From admitted to hospital to discharged from hospital,about 7 days